CLINICAL TRIAL: NCT03768284
Title: Genetic Analysis of Pediatric Psoriasis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Psoriasis Foundation (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Other Study IDs: 2018-2259
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva (or buccal swabs in the case of infants) will be obtained for DNA isolation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriasis patients: Patients (of any age) who developed psoriasis before 12 years of age and who have no family history of psoriasis in either parent.
  Interventions: Other: Saliva or buccal sample
- Parents of psoriasis patients: Parents of patients who developed psoriasis before 12 years of age
  Interventions: Other: Saliva or buccal sample
- Up to third-degree family members with or without psoriasis: Up to third-degree family members (first cousin, grandparent, great-grandparent) with or without psoriasis, if family history is indicated.
  Interventions: Other: Saliva or buccal sample

INTERVENTIONS:
Other: Saliva or buccal sample — Saliva or buccal sample

SUMMARY:
This study will ascertain approximately 150 subjects, which will include pediatric psoriasis patients diagnosed before age 12, parents not affected by psoriasis, and if a family history is indicated, up to third-degree family members. Saliva (or buccal swabs in the case of infants) will be obtained for DNA isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients (of any age) who developed psoriasis before 12 years of age and who have no family history of psoriasis in either parent.
* Parents of patients who developed psoriasis before 12 years of age
* Up to third-degree family members (first cousin, grandparent, great-grandparent) with or without psoriasis, if family history is indicated.

Exclusion Criteria:

* Patients, parents, and other family member unable to give a saliva or buccal swab sample.
* Patients, parents, and other family member unable to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will ascertain approximately 150 subjects, which will include pediatric psoriasis patients diagnosed before age 12, parents not affected by psoriasis, and if a family history is indicated, up to third-degree family members.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
CARD14 mutations | one year
  The number of pathogenic mutations identified in CARD14 in a pediatric psoriasis cohort

SECONDARY OUTCOMES:
De novo mutations | one year
  The number of candidate psoriasis genes through the identification of de novo mutations in moderate-to-severe pediatric cases who require systemic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No